CLINICAL TRIAL: NCT05856656
Title: Music Therapy as a Tool for Anxiety Reduction in Localized Breast Cancer
Acronym: CENSORIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2022-21
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Breast Cancer; Chemotherapy
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music therapy arm (Experimental): A music therapy will be offered to patients before the first 3 chemotherapy cycles
  Interventions: Behavioral: Music therapy
- Standard care arm (No Intervention): Standard patient care, no intervention

INTERVENTIONS:
Behavioral: Music therapy — Music therapy is a technique of care, accompaniment and support, which aims to improve health and well-being.
  Arms: Music therapy arm

SUMMARY:
Breast cancer is the number one cancer in women worldwide, with 58,500 new cases in metropolitan France in 2018. The announcement of the cancer, the treatment methods and their side effects can generate unpleasant emotions, such as fear, for example, and the resources for coping with them differ according to the patient. Coming to the hospital as an outpatient for chemotherapy is in itself a source of anxiety.

The use of music in the treatment process is a therapy that can help patients to reduce the intensity of their unpleasant emotions. Active music therapy involves the patient playing an instrument, including voice and body movement in rhythm, without requiring any musical skills. The presence of a qualified music therapy professional is essential, particularly in the reception of the emotions that may be generated during the sessions. These sessions can be collective or individual. In breast cancer, music therapy has been shown to be effective in reducing pain, anxiety, depressive symptoms and length of hospitalisation in patients undergoing mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with localized breast cancer
* Indication for adjuvant or neoadjuvant chemotherapy
* Patient > 18 years of age
* Patient with signed consent
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Metastatic patient
* Triple negative patient
* Patient not eligible for curative surgery
* Patient who has already received chemotherapy
* Unaided deaf patient
* Women who are pregnant, likely to be pregnant or breastfeeding
* A patient presenting a depressive episode or a psychotic pathology at the time of the initial consultation
* Patient who does not understand French
* Cognitive disorder or inability to understand,
* Patient protected by law, under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of music therapy on anxiety in breast cancer patients undergoing adjuvant or neoadjuvant chemotherapy. | 5 months
  Changes in anxiety before the first and third chemotherapy sessions will be measured using the State Trait Anxiety Inventory (= STAI etat score).

CONTACTS AND LOCATIONS:
Overall Officials: Sandra PIQUIN, Study Director — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No